CLINICAL TRIAL: NCT06033209
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of an HIV Envelope Trimer, N332-GT5 gp140, Adjuvanted With SMNP in Adult Participants Without HIV
Brief Title: A Trial to Evaluate an HIV Envelope Trimer, N332-GT5 gp140, Adjuvanted With SMNP in Adult Participants Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 144; 39021 (Other: DAIDS-ES ID)
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: The overall design of this trial involves 2 parts. In Part A, the goal is to establish the tolerability of both N332-GT5 and the SMNP adjuvant. This is a partially randomized design - Part A is nonrandomized, and Part B is randomized.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part A Intramuscular (IM) safety with dose finding - Group 1 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part A IM safety with dose finding - Group 2 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part A IM safety with dose finding - Group 3 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part A IM safety with dose finding - Group 4 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part A IM safety with dose finding - Group 5 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part A IM safety with dose finding - Group 6 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Fractioned); Biological: SMNP (IM, Fractioned)
- Part A Subcutaneous (SC) safety with dose finding - Group 7 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part A SC safety with dose finding - Group 8 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part A SC safety with dose finding - Group 9 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part A SC safety with dose finding - Group 10 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part A SC safety with dose finding - Group 11 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part A SC safety with dose finding - Group 12 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Fractioned); Biological: SMNP (SC, Fractioned)
- Part B IM Immunogenicity - Group 13 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (IM, Bolus); Biological: SMNP (IM, Bolus)
- Part B SC Immunogenicity - Group 14 (Experimental)
  Interventions: Biological: N332-GT5 gp140 (SC, Bolus); Biological: SMNP (SC, Bolus)
- Part B Immunogenicity - Group 15 (Experimental): Group 15 N332-GT5 gp140 with SMNP dose and route (SC or IM) is To Be Determined (TBD) based on groups 6 and 12 (Part A).
  Interventions: Biological: N332-GT5 gp140 (IM, Fractioned); Biological: N332-GT5 gp140 (SC, Fractioned); Biological: SMNP (IM, Fractioned); Biological: SMNP (SC, Fractioned)

INTERVENTIONS:
Biological: N332-GT5 gp140 (IM, Bolus) — IM in the deltoid
  Arms: Part A IM safety with dose finding - Group 2; Part A IM safety with dose finding - Group 3; Part A IM safety with dose finding - Group 4; Part A IM safety with dose finding - Group 5; Part A Intramuscular (IM) safety with dose finding - Group 1; Part B IM Immunogenicity - Group 13
Biological: N332-GT5 gp140 (IM, Fractioned) — IM in the deltoid, Fractionated escalating dose for prime
  Arms: Part A IM safety with dose finding - Group 6; Part B Immunogenicity - Group 15
Biological: N332-GT5 gp140 (SC, Bolus) — SC in the upper arm
  Arms: Part A SC safety with dose finding - Group 10; Part A SC safety with dose finding - Group 11; Part A SC safety with dose finding - Group 8; Part A SC safety with dose finding - Group 9; Part A Subcutaneous (SC) safety with dose finding - Group 7; Part B SC Immunogenicity - Group 14
Biological: N332-GT5 gp140 (SC, Fractioned) — SC in the upper arm, Fractionated escalating dose for prime
  Arms: Part A SC safety with dose finding - Group 12; Part B Immunogenicity - Group 15
Biological: SMNP (IM, Bolus) — IM in the deltoid
  Arms: Part A IM safety with dose finding - Group 2; Part A IM safety with dose finding - Group 3; Part A IM safety with dose finding - Group 4; Part A IM safety with dose finding - Group 5; Part A Intramuscular (IM) safety with dose finding - Group 1; Part B IM Immunogenicity - Group 13
Biological: SMNP (IM, Fractioned) — IM in the deltoid, Fractionated escalating dose for prime
  Arms: Part A IM safety with dose finding - Group 6; Part B Immunogenicity - Group 15
Biological: SMNP (SC, Bolus) — SC in the upper arm
  Arms: Part A SC safety with dose finding - Group 10; Part A SC safety with dose finding - Group 11; Part A SC safety with dose finding - Group 8; Part A SC safety with dose finding - Group 9; Part A Subcutaneous (SC) safety with dose finding - Group 7; Part B SC Immunogenicity - Group 14
Biological: SMNP (SC, Fractioned) — SC in the upper arm, Fractionated escalating dose for prime
  Arms: Part A SC safety with dose finding - Group 12; Part B Immunogenicity - Group 15

SUMMARY:
HVTN 144 is a phase 1 clinical trial to being conducted to evaluate the safety and immunogenicity of an HIV envelope trimer, N332-GT5 gp140, adjuvanted with saponin/MPLA nanoparticles (SMNP) in adult participants without HIV. The study aims to evaluate the safety and tolerability of N332-GT5 gp140 adjuvanted with SMNP in adult volunteers without HIV and in overall good health, including identifying a safe and tolerable dose, route, and schedule of administration of the novel adjuvant SMNP. The study also aims to evaluate the induction of BG18-class immunoglobulin G (IgG) B-cell responses in memory B cells by the study regimens and compare the responses between the different groups.

HVTN 144 will be conducted in 2 parts with 84 volunteers without HIV and in overall good health, aged 18 to 55 years. The study duration is 22 months which includes 8 months for enrollment, planned safety holds, follow-up, and Adverse Event of Special Interest (AESI) health contact 1 year after last vaccination.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of combining 2 FIH products: N332-GT5 gp140 HIV trimer protein adjuvanted with SMNP, co-administered as 2 bolus immunizations (week 0 and 8) or fractionated escalating dose prime (6 immunizations over 3 weeks) followed by bolus immunization boost (week 10), via either subcutaneous (SC) route in the upper arm or intramuscular (IM) route to the deltoid. N332-GT5 gp140 is based on the BG505 MD39 native-like trimer (NLT). The dose escalation study (Part A) will determine the maximum safe dose, within our schema, of N332-GT5 gp140 and SMNP for 4 vaccination modalities: IM/bolus, IM/fractionated escalating dose prime, SC/bolus, and SC/fractionated escalating dose prime. A primary endpoint will be safety and tolerability. The trial will evaluate: (1) the concept of generalized germline targeting for HCDR3-dominant bnAb precursors; (2) germline targeting for V3-glycan (V3G)-specific BG18-class bnAbs; (3) establishing a safe and effective dose of SMNP in humans; (4) immunogenicity of an HIV Env trimer adjuvanted with SMNP; and (5) ranking of HIV trimer immune response magnitude and quality for bolus/IM, bolus/SC, and fractionated escalating dose with one of either IM or SC.

ELIGIBILITY:
Inclusion Criteria:

General and demographic criteria:

1. Age of 18 through 55 years
2. Access to a participating HVTN Clinical Research Site (CRS) and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of Understanding (AoU): Volunteer demonstrates understanding of this study by completing a questionnaire prior to the first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Agrees not to enroll in another study of an investigational research agent until completion of the study
6. Good general health as shown by medical history, physical exam, and screening laboratory tests

   HIV-related criteria:
7. Willingness to receive HIV test results
8. Willingness to discuss HIV risks and amenable to HIV risk-reduction counseling
9. Assessed by the clinic staff as having a low likelihood of acquiring HIV and is committed to avoiding behaviors associated with a higher likelihood of acquiring HIV through the last required protocol clinic visit

   Laboratory inclusion values Criteria:
10. Hemoglobin (Hgb)

    * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth (AFAB)
    * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth (AMAB) and transgender men who have been on hormone therapy for more than 6 consecutive months
    * ≥ 12.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
    * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth
11. White blood cell (WBC) count = 2500 to 12000 cells/mm3 with normal differential, or differential approved by Investigator of Record (IoR) as not clinically significant
12. Total lymphocyte count ≥ 650 cells/mm3 with normal differential, or differential approved by IoR as not clinically significant
13. Remaining differential either within local lab reference range or with site physician approval
14. Platelets = 125000 to 550000 cells/mm3
15. Chemistry panel: Alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal (ULN); serum creatinine ≤ 1.1 x ULN based on the local lab reference range.
16. Corrected total serum calcium level of ≥ 8.5 mg/dL
17. Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA)
18. Negative Hepatitis B surface antigen (HBsAg)
19. Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV nucleic acid test (NAT) if the anti-HCV is positive.

    Reproductive status criteria:
20. For volunteers AFAB or intersex at birth and are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

    * Must agree to use effective means of contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment and 4 weeks after their last scheduled vaccination timepoint.
    * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) at screening (ie, prior to randomization, if applicable) and prior to study-product administration on the day of study-product administration. (Persons of pregnancy potential require a pregnancy test prior to injection 1 of the fractionated escalating dose series)
    * Persons who are NOT of pregnancy potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records) or having reached menopause (no menses for 1 year) are not required to undergo pregnancy testing.
21. AFAB volunteers or volunteers who were intersex at birth must also agree not to seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria:

General criteria:

1. Blood products received within 120 days before first vaccination
2. Investigational research agents received within 30 days before first vaccination
3. Body mass index (BMI) ≥ 40, or BMI ≥ 35 with 2 or more of the following: Age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
4. Intent to participate in any other study that requires non-HVTN HIV Ab testing during the planned duration of the HVTN 144 study
5. Pregnant or breastfeeding
6. Active duty and reserve US military personnel

   Vaccines and other injections criteria:
7. HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 144 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
8. Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational. Exceptions may be made by the HVTN 144 PSRT on a case-by-case basis.
9. Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 144 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 144 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) more than 1 year ago, eligibility for enrollment will be determined by the HVTN 144 PSRT on a case-by-case basis.
10. Live attenuated vaccines received within 30 days before the first vaccination or scheduled within 28 days after injection (eg, measles, mumps, and rubella (MMR); oral polio vaccine (OPV); varicella; yellow fever; live attenuated influenza vaccine). ACAM2000 vaccine >28 days prior with a vaccination scab still present.
11. Any vaccines that are not live attenuated vaccines and were received within 14 days prior to the first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B). Please note this includes incompetent vaccine such as the Jynneos vaccine for the prevention of mpox disease.
12. Allergy treatment with antigen injections within 30 days before the first vaccination or that are scheduled within 14 days after the first vaccination

    Immune system criteria:
13. Immunosuppressive medications received within 168 days before first vaccination (not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment)
14. Serious adverse reactions to vaccines or to vaccine components such as AS01B ("Shingrix") or Matrix M (Novovax CoV2373), including history of anaphylaxis and related symptoms, such as hives, respiratory difficulty, angioedema, and/or abdominal pain (not exclusionary: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child).
15. IgG received within 60 days before first vaccination (for mAbs, see criterion #8 above)
16. Autoimmune disease, current or history (not exclusionary: mild, well-controlled psoriasis)
17. AESIs: Volunteers who currently have, or have a history of, any condition that could be considered an AESI for the product(s) administered in this protocol.
18. Immunodeficiency

    Clinically significant medical conditions criteria:
19. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated injections or blood draws,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
    * Any condition specifically listed among the exclusion criteria below.
20. Any medical, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
21. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
22. Current anti-tuberculosis (TB) prophylaxis or therapy
23. Asthma exclusion criteria:

    Asthma is excluded if the participant has ANY of the following:
    * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium- to high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent) or more than 1 medication for maintenance therapy daily. For example, potential participants taking long-acting bronchodilator/inhaled corticosteroid combinations for daily maintenance are excluded (note: maintenance monotherapy with cromolyn, leukotriene receptor antagonist, or theophylline is not exclusionary).
24. Diabetes mellitus type 1 or type 2 (not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes)
25. Thyroidectomy, or thyroid disease requiring medication during the last 12 months (not exclusionary: well-controlled non-autoimmune thyroid disease)
26. Hypertension: The average systolic blood pressure between the screening visit and the enrollment visit must be below 140 mmHg. The average diastolic blood pressure between the screening visit and the enrollment visit must be below 90 mmHg. A single measurement greater than or equal to 160 mmHg systolic or 100 mmHg diastolic during the current study evaluation is exclusionary.
27. Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
28. Malignancy (not exclusionary: volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
29. Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
30. Asplenia: Any condition resulting in the absence of a functional spleen
31. History of angioedema or anaphylaxis (not exclusionary: angioedema or anaphylaxis with known trigger and no episodes within 5 years)
32. History of generalized urticaria within past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms (solicited adverse events) will be collected | Through study completion, an average of 1 year
Systemic reactogenicity signs and symptoms (solicited adverse events) will be collected | Through study completion, an average of 1 year
Number of Serious Adverse Events (SAEs) leading to early participant withdrawal or permanent discontinuation | 35 weeks and for 12 months following any receipt of study product
Number of Medically attended adverse events (MAAEs) leading to early participant withdrawal or permanent discontinuation | 35 weeks and for 12 months following any receipt of study product
Number of AESIs leading to early participant withdrawal or permanent discontinuation | 35 weeks and for 12 months following any receipt of study product
Number of Adverse Events (AEs) leading to early participant withdrawal or permanent discontinuation | 35 weeks and for 12 months following any receipt of study product
Comparison of number of reported/assessed local and systemic reactogenicity, SAE's and AESI's and medically attended adverse events at increasing doses of adjuvant at constant dose of N332-GT5 gp140 | 35 weeks
Frequency of BG18 epitope-specific B cells as determined by flow cytometry | 35 weeks
Proportion of participants with BG18-class IgG memory B cells in peripheral blood mononuclear cell (PBMCs), measured by antigen-specific B-cell sorting, B-cell receptor (BCR) sequencing, and bioinformatic analysis | 35 weeks
Frequency of BG18-class B cells among IgG memory B cells in PBMCs, measured by antigen-specific B-cell sorting, BCR sequencing, and bioinformatic analysis | 35 weeks

SECONDARY OUTCOMES:
Proportion of participants with BG18-class IgG B cells, measured by antigen-specific B-cell sorting, BCR sequencing, and bioinformatic analysis | 35 weeks
Frequency of BG18-class B cells among IgG B cells in germinal centers (GCs), measured by antigen-specific B-cell sorting, BCR sequencing, and bioinformatic analysis | 35 weeks
Response rate of serum binding Ab responses to N332-GT5 gp140 and BG18 epitope on the trimer measured by binding antibody multiplex assay (BAMA) | 35 weeks
Magnitude of serum binding Ab responses to N332-GT5 gp140 and BG18 epitope on the trimer measured by binding antibody multiplex assay (BAMA) | 35 weeks
Response rate of serum neutralizing antibodies (nAbs) that neutralize pseudoviruses engineered to be sensitive to BG18-precursors | 35 weeks
Concentration of serum nAbs that neutralize pseudoviruses engineered to be sensitive to BG18-precursors | 35 weeks
Frequency of N332-GT5 gp140 trimer-specific B cells | 35 weeks
Frequency of BG18 sequences isolated postvaccination | 35 weeks
Magnitude of binding Abs measured by BAMA | 35 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital
Locations (8):
- United States (8):
  - Bridge HIV CRS, San Francisco, California
  - Atlanta - Hope Clinic, Decatur, Georgia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - New York Blood Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Penn Prevention CRS [Site ID: 30310], Philadelphia, Pennsylvania
  - Vanderbilt Institute for Infection, Immunology and Inflammation, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No